CLINICAL TRIAL: NCT02411188
Title: For Her Heart's Sake: A Clinical Trial to Assess Strategies to Enhance Participation in Cardiac Rehabilitation - STEP Project
Brief Title: For Her Heart's Sake STEP Project: A Clinical Trial
Acronym: FHHS: STEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues; changed protocol to prospective cohort study
Sponsor: University of Manitoba (Other)
Collaborators: Victoria General Hospital Foundation (Unknown); Reh-Fit Fitness Centre (Unknown); Wellness Institute-Seven Oaks General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UManitoba
Record Dates: First submitted 2015-03-30; First posted 2015-04-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2015-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STEP Program Group (Experimental): Arm: Intervention: The 12-week STEP Program intervention will include: initial individual consult/goal setting; weekly 90 minute information/interactive sessions; individualized patient centred care; journaling
  Interventions: Behavioral: The STEP Program
- Usual Care Group (No Intervention): The usual care group will follow the routine model of care for post-discharge patients who do not participate in a CRP. Usual care group participants will be given the opportunity/option to participate in the STEP Program in 6 months.

INTERVENTIONS:
Behavioral: The STEP Program — Intervention: The 12-week STEP Program will include: initial individual consult/goal setting; weekly 90 minute information/interactive sessions; individualized patient centred care; journaling
  Arms: STEP Program Group

SUMMARY:
The goal of the proposed project is to determine if providing an intervention for women who decline the invitation to participate in standard cardiac rehabilitation programs (CRPs) will ultimately result in an increase their participation in CRPs.This study will evaluate outcomes of patients randomized to the FHHS STEP Program versus by non-STEP Program participants. The overall goal is to provide an alternate, introductory program that will engage, educate, and empower women following a cardiac event. Providing these women with the necessary personal resources will encourage and enable these women to take the step towards a cardiac rehabilitation program, which, in turn will ideally lead to a life-long commitment to heart health.

DETAILED DESCRIPTION:
Cardiac rehabilitation programs (CRPs) have been shown to improve outcomes following a cardiac event. Referrals to the CRP are a standard part of the community-based continuing care process within the Winnipeg region, to include automatic referrals for hospitalized patients, based on specific criteria, physician referrals and self-referrals. However, fewer women than men are referred to and participate in CRPs in Winnipeg.

The investigators' study is unique in that the investigators plan to capture those women who may not be ready to change or participate in a traditional CRP. While women who are in the pre-contemplative or contemplative stages of change may not be ready to participate in a standard CRP, they may be willing to explore a complementary opportunity: the FHHS STEP Program. The overall goal of this project is to provide a collaborative team environment that will engage women; educate, and empower women; and provide women with the necessary personal resources to enable them to take the step towards a cardiac rehabilitation program and a life-long commitment to heart health. The investigators' 2-group randomized clinical trial will compare physiological and psychosocial outcomes among women completing a 12-week gender specific introduction to cardiac rehabilitation with non-program attenders.

ELIGIBILITY:
Inclusion Criteria:

* Discharged from a Winnipeg Regional Health Authority (WRHA) facility;
* Diagnosis of stable ischemic heart disease or acute coronary syndrome who have undergone revascularization via coronary artery bypass graft (CABG) surgery or elective percutaneous coronary intervention (PCI);
* Diagnosis of valvular heart disease who have undergone valve surgery;
* Diagnosis of stable ischemic or non-ischemic heart failure;
* Able to read, write, and speak English;
* Referred to and declined participation in a CRP in Winnipeg;
* Willing and able to attend the STEP Program at the Victoria General Hospital.

Exclusion Criteria:

* Patients who have unstable or recent unstable cardiac syndrome, as defined by:

  * Severe heart failure (New York Heart Association Class IV) or angina (Canadian Cardiovascular Society Class IV) symptoms
  * Non-re-vascularized > triple vessel disease
* Non-repaired severe valvular heart disease (aortic or mitral area < 1.0cm2 or mean gradient > 40 mmhg or > 10mmHg [millimetres of mercury] respectively)
* Severe systolic heart failure (LVEF [left ventricular ejection fraction] < 30%)
* High risk stress test
* Exercise induced ventricular arrhythmias or recent (within the past 6 months) hospitalization for ventricular arrhythmias
* Unstable arrhythmias (i.e., bradycardia; tachyarrhythmias)
* Previous attendance in a CRP
* Physical limitations that would preclude ability to walk
* Cognitive impairment/deficits that would preclude participation in the STEP Project
* Automatic internal cardiac defibrillator in situ
* On waitlist for cardiac procedure (e.g., cardiac surgery; PCI)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Cardiac Rehabilitation Program Enrolment | 12 months
  3 yes/no questions: have you contacted a CRP; have you joined a CRP; do you plan to contact a CRP. if not, why not

SECONDARY OUTCOMES:
Short-Form-36 | baseline, 3, 6 and 12 months
  36 items re 8 dimensions: physical functioning (10 items), role limitations - physical (4 items), bodily pain (2 items), social functioning (2 items), general mental health (5 items), role limitations - emotional (3 items), vitality (4 items), general health perceptions, 5 items); coded to 0-100 score, with higher values representing more favourable states
Brief Symptom Inventory | baseline, 3, 6 and 12 months
  53 items; 5-point Likert scale (1-5); operationalizes concepts of anxiety, depression and hostility; 9 symptom domains, with higher scores indicating greater levels of distress.
General Self-Efficacy Scale | baseline, 3, 6, 12 months
  10 items; scoring based on 4-point Likert scale (1-4), with higher scores reflecting higher perceived self-efficacy
Multidimensional Self-Efficacy for Exercise Scale | baseline, 3, 6 and 12 months
  9 items; 11-point Likert scale (0-10), with higher scores reflecting higher task efficacy (3 items), coping efficacy (3 items) and scheduling efficacy (3 items
Enhancing Recovery in Coronary Heart Disease Social Support Instrument | baseline, 3, 6 and 12 months
  7 item scale is scored by totalling the six 5-point Likert scale items and a 7th item, which is scored 4 for 'yes' and 2 for 'no'. The scale captures structural, emotional and instrumental support
Stages of Change Questionnaire | baseline, 3, 6 and 12 months
  12 5-point-Likert scale (1-5) questions; Stages of readiness to change for each of the listed behaviors include 5 response items representing each of the stages of change (i.e., precontemplation, contemplation, preparation, action, and maintenance).
Health Resource Utilization Questionnaire | 3, 6 and 12 months
  4-items: self-reported number of contacts/visits with primary care provider, cardiologist, emergency department/Walk-in Clinic visits and hospital admissions.
International Physical Activity Questionnaire | baseline, 3, 6 and 12 months
  9-item, subjective 7 day recall of physical activity patterns
Client Satisfaction Questionnaire | 3 months
  intervention group only; 8 items; 4-point Likert scale; assesses general satisfaction with the health care services received; higher scores reflect higher satisfaction
6-Minute Walk Test | baseline, 3, 6 and 12 months
  total distanced walked in 6 minutes
Accelerometry | baseline, 3, 6 and 12 months
  accelerometers monitor/measure physical activity/sedentary behaviours for a specified period of time (7 days).

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Ann V Sawatzky, RN, PhD, Principal Investigator — University of Manitoba